CLINICAL TRIAL: NCT06493604
Title: A Randomized, Double-Masked, Vehicle-Controlled Parallel Group Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: A Trial to Assess the Safety and Efficacy of Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADX-102-DED-032
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye Disease
Keywords: reproxalap
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%)
- Vehicle Ophthalmic Solution administered six times over two consecutive days (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) — Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days
  Arms: Reproxalap Ophthalmic Solution (0.25%) administered six times over two consecutive days
Drug: Vehicle Ophthalmic Solution — Vehicle Ophthalmic Solution administered six times over two consecutive days
  Arms: Vehicle Ophthalmic Solution administered six times over two consecutive days

SUMMARY:
A Randomized, Double-Masked, Vehicle-Controlled Parallel Group Clinical Trial to Assess Efficacy and Safety of 0.25% Reproxalap Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

DETAILED DESCRIPTION:
Dry eye chamber challenge trial

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age (either gender and any race)
* Ability to provide written informed consent and sign the Health Information Portability and Accountability Act form
* Reported history of ocular discomfort associated with dry eye disease for at least 6 months prior to Visit 1
* Reported history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* Clinically significant slit lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters
* Diagnosis of an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1
* Contact lens use within 7 days of Visit 1 or anticipated use of contact lenses during the trial
* Previous laser-assisted in situ keratomileusis surgery within the last 12 months
* Systemic corticosteroid or other immunomodulator therapy (not including inhaled corticosteroids) within 14 days of Visit 1, or any planned immunomodulatory therapy throughout the clinical trial
* Use of and unwillingness to discontinue topical ophthalmic prescriptions (including medications for glaucoma) or over-the-counter solutions (not including artificial tears), gels, or scrubs for the duration of the trial (excluding medications allowed for the conduct of the trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Ocular discomfort symptom score over 100 minutes in the dry eye chamber at Visit 1 and Visit 3 | Day -14 to Day 2
  Measured using a 0 - 100 visual analog scale (VAS) where 0 is "no discomfort" and 100 is "maximal discomfort"

CONTACTS AND LOCATIONS:
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT06493604/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT06493604/SAP_001.pdf